CLINICAL TRIAL: NCT04677894
Title: Comparison of Video Laryngoscopy and Direct Laryngoscopy for Nasotracheal Intubation During Pediatric Dental Surgery: a Randomized Clinical Trial
Brief Title: Comparison of Video Laryngoscopy and Direct Laryngoscopy for Nasotracheal Intubation During Pediatric Dental Surgery
Acronym: Laryngoscopy
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Ebru Canakci, M.D.,Associated Professor ,Head of Department of Anesthesiology and Reanimation, Ordu University
Other Study IDs: ECanakci
Record Dates: First submitted 2020-11-29; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Airway Complication of Anesthesia; Peroperative Complication; Intraoperative Hypertension; Tachycardia, Sinus; Desaturation of Blood
Keywords: pediatric oral surgery; direct laryngoscopy; video laryngoscopy; nasotracheal intubation
MeSH Terms: conditions — Intraoperative Complications; Tachycardia, Sinus | interventions — Laryngoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Direct Laringoscopy: Group DL: Group of patients intubated using a Macintoch blade laryngoscope.
  Interventions: Device: Laryngoscopy
- Group Videolaringoscopy: Group VL: Group of patients intubated using a McGrath video laryngoscope.
  Interventions: Device: Laryngoscopy

INTERVENTIONS:
Device: Laryngoscopy — During the intubation, the head of the patient was kept in a neutral position, patients were nasotracheally intubated

SUMMARY:
Background and Objective: Airway control is a condition that should be evaluated primarily in anesthesia practice in the pediatric age group. Failed intubation or prolonged intubation duration can cause atelectasis and hypoxia in children. The aim of this study was to examine the effects of Macintosh laryngoscopy and McGrath videolaryngoscopy on hemodynamic parameters in pediatric patients who were scheduled to undergo elective dental surgery and required intubation for the application of general anesthesia.

Methods: Sixty-six patients were divided into two groups according to the procedure used during intubation, namely, direct laryngoscopy or video laryngoscopy. The Cormack-Lehane and Mallampati scores, intubation duration, heart rate at minutes 0, 1, 3 and 5 during intubation, mean arterial pressure, EtCO2and SpO2 values were recorded for all the patients.

DETAILED DESCRIPTION:
Many techniques in the management of a difficult airway have been used in adult patients. In pediatric patients, awake fiberoptic intubation is difficult or even impossible . The video laryngoscope is a new tool produced by combining video technology and laryngoscope. Published studies on the video laryngoscope were mostly performed in adults . In this study, we used a Macintosh laryngoscope, which is a routinely used tool in anesthesiology, and a McGrath video laryngoscope, which is a type of a newly developed video laryngoscope that has not widely been used in the pediatric age group. The aim of this study was to examine the effects of Macintosh laryngoscopy and McGrath videolaryngoscopy on hemodynamic parameters in pediatric patients who were scheduled to undergo elective dental surgery and required intubation for the application of general anesthesia. We also evaluated whether Macintosh laryngoscopy and McGrath videolaryngoscopy improved the stress response and whether these approaches facilitated the intubation procedure.

ELIGIBILITY:
Inclusion Criteria:

Healthy children between the ages of 4-13

* Ordu University School of Medicine ,pediatric age group ,elective oral surgery 4-13 years and who were scheduled for elective oral surgery under general anesthesia with intubation If Patients with a Cormack -Lehane score 1,2 or 3 and if Mallampathy score of 1,2 or 3 were inccluded from the study

Exclusion Criteria:

1. With malignancy disease patients
2. with norological disorders
3. with congenital heart disease
4. with airway abnormality
5. with airway disease patients
6. Patients age Under 4 years , Above 13 years
7. If Patients with a Cormack -Lehane score 4 and if Mallampathy score of 4 were excluded from the study -

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study included 66 ASA I-II patients with an age range of 4-13 years and who were scheduled for elective dental surgery under general anesthesia with intubation.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate | During surgery 0. minute
  Heart Rate (HR)
Heart Rate | During surgery 1. minute
  Heart Rate (HR)
Heart Rate | During surgery 3. minute
  Heart Rate (HR)
Heart Rate | During surgery 5. minute
  Heart Rate (HR)
Heart Rate | During surgery 10. minute
  Heart Rate (HR)
Mean Arterial Pressure | During surgery 0. minute
  Mean Arterial Pressure (MAP)
Mean Arterial Pressure | During surgery 1. minute
  Mean Arterial Pressure (MAP)
Mean Arterial Pressure | During surgery 3. minute
  Mean Arterial Pressure (MAP)
Mean Arterial Pressure | During surgery 5. minute
  Mean Arterial Pressure (MAP)
Mean Arterial Pressure | During surgery 10. minute
  Mean Arterial Pressure (MAP)
Saturation | During surgery 0. minute
  SpO2
Saturation | During surgery 1. minute
  SpO2
Saturation | During surgery 3. minute
  SpO2
Saturation | During surgery 5. minute
  SpO2
Saturation | During surgery 10. minute
  SpO2
End Tidal Carbondioxide | During surgery 0. minute
  EtCO2
End Tidal Carbondioxide | During surgery 1. minute
  EtCO2
End Tidal Carbondioxide | During surgery 3. minute
  EtCO2
End Tidal Carbondioxide | During surgery 5. minute
  EtCO2
End Tidal Carbondioxide | During surgery 10. minute
  EtCO2

SECONDARY OUTCOMES:
Entubation Time | During Surgery 1.minute
  Entubation time , (minute)
Entubation Time | During Surgery 2.minute
  Entubation time , (minute)
Entubation Time | During Surgery 3.minute
  Entubation time , (minute)

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Canakci, MD, Principal Investigator — Ordu University School of Medicine Department of Anesthesiology and Reanimation; Ahmet Gultekin, MD, Study Chair — Namık Kemal University School of Medicine Department of Anesthesiology and Reanimation
Locations (1):
- Ordu University School of Medicine ,Department of Anesthesiology and Reanimation, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No